CLINICAL TRIAL: NCT01791907
Title: Effect of Structured Education in Advanced Carbohydrate Counting or Healthy Food Choices With Low Glycemic Index in Type 1 Diabetes
Brief Title: Effect of Structured Nutrition Education in Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPN 304-12
Record Dates: First submitted 2013-02-07; First posted 2013-02-15 (Estimated); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

ARMS (3):
- Structured education in carbohydrate counting (Experimental): A structured education in carbohydrate counting, a course inspired by the DAFNE program (Dose Adjustment For Normal Eating)
  Interventions: Behavioral: Structured education in carbohydrate counting
- Structured education in healthy food choices and low GI (Experimental): A new, structured education for heart healthy food choices and low glycemic index in type 1 diabetes. The education is called "My Wellness-LADDER" (Lifelong Adult Diet & Diabetes Education Resource) and it is specifically designed to provide high long-term adherence through improved empowerment and transformative life style change.
  Interventions: Behavioral: Structured education in healthy food choices and low glycemic index
- Regular routine (No Intervention)

INTERVENTIONS:
Behavioral: Structured education in carbohydrate counting
  Arms: Structured education in carbohydrate counting
Behavioral: Structured education in healthy food choices and low glycemic index
  Arms: Structured education in healthy food choices and low GI

SUMMARY:
Type 1 diabetes (T1DM) is a chronic disease that affects approximately 10% of all diabetes patients in the world. Diabetes a serious disease in which life expectancy is reduced, largely due to increased mortality from kidney disease and cardiovascular (CVD) disease. Poor glycemic control also results in eye and nerve damage, and psychosocial stress. Good metabolic control, e.g. normalized hemoglobin levels (HbA1c) and normal blood lipids, reduces the risk of eye, kidney, nerve, and vascular damage. Proper nutrition can normalize blood sugar levels, improve blood lipids and prolong life in people with diabetes, according to Swedish Council on Health Technology Assessment (SBU).

Dietary treatment is therefore seen as pivotal in the treatment of diabetes. This project aims to evaluate two methods of structured training in patients with type 1 diabetes:

1. A structured education in carbohydrate counting, a course inspired by the DAFNE program (Dose Adjustment For Normal Eating)
2. A new, structured education for heart healthy food choices and low glycemic index in type 1 diabetes. The education is called "My Wellness-LADDER" (Lifelong Adult Diet & Diabetes Education Resource) and it is specifically designed to provide high long-term adherence through improved empowerment and transformative life style change.

The methods are compared with regular routine (control group).

This is a randomized controlled trial with three intervention groups 1) Healthy food choices with a low glycemic index, 2) carbohydrate counting, and 3) regular routine. Follow-up period is 1 year. Eight Swedish specialist clinics are participating and 24 patients at each clinic are to be enrolled.

The hypotheses is that structured group education on heart healthy food choices and low glycemic index provide the same improvement in glycemic control and quality of life as advanced carbohydrate counting in T1DM, as compared to regular routine. An additional hypotheses is that structured education on healthy food choices and low glycemic index leads to larger CVD risk factor reductions in T1DM compared to carbohydrate counting and regular routine and that structured education on healthy food choices and low glycemic index lead to more heart healthy food choices in T1DM compared to carbohydrate counting and regular routine. Lastly, the hypotheses is that structured education on healthy food choices and low glycemic index lead is more cost effective in T1DM compared to carbohydrate counting and regular routine.

ELIGIBILITY:
Inclusion Criteria:

* Having type 1 diabetes
* Diabetes duration > 3 years
* Age 20-70 years
* BMI <35 (kg/m2)
* Multiple dose injection (MDI) therapy
* HbA1c 57-78 mmol/mol
* Being healthy other than diabetes
* Autonomous accommodation and having influence over one's own food choices.
* Have given informed consent to participate in the study, as well as having the ability of oral and written communication in Swedish.

Exclusion Criteria:

* Nephropathy (dU albumin> 300 mg / d)
* Retinopathy (grade> 2)
* Foot ulcers
* Gastroparesis
* Difficulties visiting the hospital
* Current or planned pregnancy during the study period
* ≥ 14 days fast during the study period
* Having partaken in education in carbohydrate counting (≥ 4 hours) in the last two years
* No computer access

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
HbA1c | 1 year
  The primary outcome measure is to detect a clinically significant difference in HbA1c (= 4.2 mmol / mol) between the three treatment arms

SECONDARY OUTCOMES:
Quality of life | 1 year
  Secondary measures is to demonstrate a difference between the groups in terms of quality of life
CVD risk factors | 1 year
  Secondary measures is to demonstrate a difference between the groups in terms of CVD risk factors
Hypoglycemia | 1 year
  Secondary objectives is to demonstrate a difference between the groups in terms of hypoglycemia
Food choices | 1 year
  To demonstrate a difference between the groups in terms of food choices
Health economics | 1 year
  A secondary objective is to demonstrate a difference between the groups in terms of health economics and compare cost- effectiveness of the treatment arms

CONTACTS AND LOCATIONS:
Overall Officials: Mette Axelsen, PhD, Principal Investigator — Göteborg University